CLINICAL TRIAL: NCT00474825
Title: Phase I Clinical Trial of Hyperbaric Oxygen Combined With Radiation and Chemotherapy for Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Dose Escalation Study of Hyperbaric Oxygen With Radiation and Chemotherapy to Treat Squamous Cell Carcinoma of the Head and Neck
Acronym: HBO-XRT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Baromedical Services (Other)
Collaborators: Prisma Health-Midlands (Other); Mayo Clinic (Other); Dartmouth-Hitchcock Medical Center (Other); Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Dick Clarke, President, National Baromedical Research Foundation, National Baromedical Services
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRF 06-01; ISRCTN12244200
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Carcinoma, Squamous Cell; Cancer of the Head and Neck
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Hyperbaric Oxygen twice weekly (Monday & Friday) with Radiation and Chemotherapy
  Interventions: Drug: Hyperbaric Oxygen Therapy; Drug: Hyperbaric Oxygen
- 2 (Active Comparator): Hyperbaric Oxygen three times per week (Monday, Wednesday & Friday) with Radiation and Chemotherapy.
  Interventions: Drug: Hyperbaric Oxygen Therapy; Drug: Hyperbaric oxygen
- 3 (Active Comparator): Hyperbaric Oxygen Five times per week (Monday through Friday) with Radiation and Chemotherapy
  Interventions: Drug: Hyperbaric Oxygen Therapy; Drug: Hyperbaric oxygen

INTERVENTIONS:
Drug: Hyperbaric Oxygen Therapy — Compression rate (breathing oxygen): per patient tolerance; 1 - 3 psi per minute Treatment dose: 2.4 ATA oxygen Treatment period: 30 minutes at 2.4 ATA Decompression rate (breathing oxygen): 2 - 3 psi per minute
Drug: Hyperbaric Oxygen — Compression rate (breathing oxygen): per patient tolerance; 1 - 3 psi per minute Treatment dose: 2.4 ATA oxygen Treatment period: 30 minutes at 2.4 ATA Decompression rate (breathing oxygen): 2 - 3 psi per minute
  Arms: 1
Drug: Hyperbaric oxygen — Compression rate (breathing oxygen): per patient tolerance; 1 - 3 psi per minute Treatment dose: 2.4 ATA oxygen Treatment period: 30 minutes at 2.4 ATA Decompression rate (breathing oxygen): 2 - 3 psi per minute
  Arms: 2
Drug: Hyperbaric oxygen — Compression rate (breathing oxygen): per patient tolerance; 1 - 3 psi per minute Treatment dose: 2.4 ATA oxygen Treatment period: 30 minutes at 2.4 ATA Decompression rate (breathing oxygen): 2 - 3 psi per minute
  Arms: 3

SUMMARY:
This research is being done because we do not know the best treatment for advanced Squamous Cell Carcinoma of the Head and Neck. These cancers have been treated with a combination of surgery, radiation and chemotherapy in varying combination. When the tumor is inoperable, radiation therapy is used with or without chemotherapy in the hope of curing the tumor.

Recently, it has become recognized as generalized knowledge that cancer cells are hypoxic (low oxygen concentration). Because of the low oxygen concentrations, many cancer treatments have not been successful. The theory behind this study is to give oxygen to patients prior to chemotherapy and radiation in hopes of generating greater results in killing cancer cells. The purpose of this study has two main objectives. The primary objective is to determine patient tolerance to each arm of the trial.

The second objective is to determine the feasibility of treatment delivery and acute toxicities associated with each regimen.

It is our intention to undertake a randomized and controlled trial should this Phase I trial prove successful in terms of patient tolerance.

DETAILED DESCRIPTION:
The goal of this study is to see if patients can tolerate HBO therapy up to five days a week.

Three patients in Arm 1 (HBO on Monday and Friday) will be observed throughout their course of concomitant radiation, chemo and hyperbaric therapy. If these patients appear to tolerate this protocol well, and no adverse effects that can be directly attributed to HBO are observed, then three more patients will be recruited for Arm 2 (HBO on Monday, Wednesday, and Friday). If again these patients appear to tolerate this protocol well, and no adverse effects that can be directly attributed to HBO are observed, then a third group of three patients will be recruited for Arm 3 (HBO Monday through Friday).

If Grade IV acute toxicity is reported for a single patient in any of the arms, 3 more patients will be recruited in the same arm. If no further adverse events occur, the protocol progresses to the next arm. If Grade IV acute toxicity is observed even a single patient, the study will be stopped.

Tumor and/or lymphatic tissue specimens will be obtained prior to starting treatment. Tumor tissue specimens will be analyzed to determine whether there is a predictive susceptibility of tumors to HBO sensitization using currently defined biomarkers known to correlate with survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological proof (from the primary lesion and/or lymph nodes) of squamous cell carcinoma of the oral cavity, oropharynx, or hypopharynx.
* Patients should have Stage III or IV disease, M0
* Patients must have life expectancy of at least 6 months and a Karnofsky performance status of ≥ 70
* Age ≥ 18 years and ≤ 70 years
* No distant metastatic disease
* No clinically significant heart disease:
* No significant ventricular arrhythmia requiring medication with antiarrhythmics
* No symptomatic coronary artery disease (angina)
* No myocardial infarction within the last 6 months
* No second or third degree heart block or bundle branch block or clinically significant conduction system abnormality
* Patients must sign a study-specific informed consent form

Exclusion Criteria:

* Histology other than squamous cell carcinoma
* Evidence of metastasis (below the clavicle or distant) by clinical or radiographic means
* Prior complete resection of the primary tumor
* Prior chemotherapy (Bleomycin) for head and neck cancer or radiotherapy to the head and neck
* Patients with simultaneous primaries
* Pregnancy
* Pulmonary pathologies (risk of decompression-induced pulmonary barotrauma):
* Current, untreated pneumothorax
* Previous history of pneumothorax
* Previous history of intrathoracic surgery
* History of pulmonary blebs or bullous lung disease
* Associated with CO2 retention
* Poorly controlled or associated with acute bronchospasm
* Where the hyperbaric physician deems the patient to have an unacceptable risk for hyperbaric treatments
* Claustrophobia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Patient tolerance to each arm of the study | During intervention phase

SECONDARY OUTCOMES:
Grade IV acute toxicities associated with each arm of the study | During intervention phase

CONTACTS AND LOCATIONS:
Overall Officials: Dick Clarke, CHT, Study Director — The Baromedical Research Foundation; Surjeet S Pohar, MD, Principal Investigator — Eastern Virginia Medical School / Norfolk General Hospital; Jay Buckey, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Robert Foote, MD, Principal Investigator — The Mayo Clinic
Locations (3):
- United States (3):
  - The Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Norfolk General Hospital / Eastern Virginia Medical School, Norfolk, Virginia

REFERENCES:
- [Background] Hartford AC, Davis TH, Buckey JC, Foote RL, Sinesi MS, Williams BB, Fariss AK, Schaner PE, Claus PL, Okuno SH, Hussey JR, Clarke RE. Hyperbaric Oxygen as Radiation Sensitizer for Locally Advanced Squamous Cell Carcinoma of the Oropharynx: A Phase 1 Dose-Escalation Study. Int J Radiat Oncol Biol Phys. 2017 Mar 1;97(3):481-486. doi: 10.1016/j.ijrobp.2016.10.048. Epub 2016 Nov 15. PMID 28126298